CLINICAL TRIAL: NCT02361606
Title: An Internet Cognitive-Behavioral Intervention for Youth With Type 1 Diabetes - Participation and Efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Orit Hamiel (Other Government)
Collaborators: Academic College of Tel Aviv-Jaffa (Other); Maccabi Healthcare Services, Israel (Other)
Responsible Party: Sponsor-Investigator, Dr. Orit Hamiel, Specialist in Pediatric Endocrinology, Pediatric Endocrinology and Juvenile Deibetes Head Department, Sheba Medical Center; Head of Juvenile Diabetes Center, Maccabi Health Services, Sheba Medical Center
Organization: Sheba Medical Center (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2009108
Record Dates: First submitted 2015-02-03; First posted 2015-02-12 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Type 1 Diabetes
Keywords: adolescents; cognitive behavioral internet intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Internet CBT intervention (Experimental): Eligible candidates were offered to participate in an internet cognitive behavioral intervention.
  Interventions: Behavioral: An Internet Cognitive-Behavioral Intervention

INTERVENTIONS:
Behavioral: An Internet Cognitive-Behavioral Intervention — We developed a cognitive behavioral program for adolescents with type 1 Diabetes and their parents, that consists of six virtual sessions at https://minustress.com/diabetes/gate.asp.
  Other Names: Minustress For Type 1 Diabetes Program; An Internet CBT for Youth with Type 1 Diabetes

SUMMARY:
Adolescents are often reluctant to receive psychological help. The investigators developed a web-based cognitive behavioral self-help intervention for adolescents with type 1 diabetes. The investigators aimed to examine the participation rate and outcomes on glycemic control and quality of life.

DETAILED DESCRIPTION:
Adolescents are often reluctant to receive psychological help. The investigators developed a web-based cognitive behavioral self-help intervention for adolescents with type 1 diabetes. The investigators aimed to examine the participation rate and outcomes on glycemic control and quality of life.

Single center study was conducted to describe participation and efficacy of internet cognitive-behavioral intervention for youth with type 1 diabetes. Adolescents with type 1 diabetes, aged 13-20 years, treated at a Juvenile Diabetes Center, were offered to participate in the intervention. Recruitment period lasted for 2 months, during January-February, 2011.

HbA1c measures of adolescents that agreed to participate, were obtained from medical records.The adolescents, that logged in, were asked to complete questionnaires before the intervention assessing their expectations of the program, quality of life and parental support. After completion of questionnaires, the adolescents were encouraged to complete 6 virtual sessions. Satisfaction was assessed after each session. In the end of the program, participants were asked again to complete questionnaires. HbA1c levels were obtained again for participants that logged in, and for participants that passively refused, 3 months or more after the recruitment.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis with diabetes for at least 1 year
* treated at Juvenile Diabetes Center
* fluent Hebrew speakers

Exclusion Criteria:

* no previous diagnosis of a psychiatric condition (such as an eating disorder)
* no opposition to the internet due to religious issues.

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 89 (Actual)
Dates: Start 2009-03; Primary Completion 2011-02 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change in quality of life. (Diabetes Quality of Life (DQOL) questionnaire) | Change from baseline to the end of intervention (3 to 6 months from baseline)
  Filled in the intervention website.
Perceived parent support. (Short version of the Social Provision Scale) | Change from baseline to the end of intervention (3 to 6 monts)
  Short version of the Social Provision Scale -filled in the intervention website.
Youth satisfaction of the program. (Questionnaire regarding the degree that the session was helpful.) | Measured at the end of every virtual session (2 days to 6 months from baseline).
  Questionnaire regarding the degree that the session was helpful.

SECONDARY OUTCOMES:
Change in glycemic control. (HbaA1c levels, obtained from medical records) | Last HbA1C before recruitment period and first HbA1C after recruitment period were obtained from medical records (3-12 months from baseline).
  HbaA1c levels, obtained from medical records twice - the closest measurement available before the trial period, and closest measurement available 3 months or more after the trial period.

OTHER OUTCOMES:
Youth expectations of the program. (Questionnaire regarding the expectations of the possible benefits of the program.) | Baseline
  Questionnaire regarding the expectations of the possible benefits of the program.

CONTACTS AND LOCATIONS:
Overall Officials: Orit Pinhas Hamiel, MD, Study Director — Sheba Medical Center; Daniel Hamiel, PhD, Study Director — The Interdisciplinary Center; Irena Vusiker, MA, Principal Investigator — Sheba Medical Center